CLINICAL TRIAL: NCT01312129
Title: Effects of Sulfasalazine on BOLD Response to Alcohol Cues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Mind Research Network (Other)
Responsible Party: Principal Investigator, Kent Hutchison, Ph.D., Professor of Translational Research, The Mind Research Network
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-381
Record Dates: First submitted 2011-03-09; First posted 2011-03-10 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Alcohol Dependence
Keywords: Alcohol; Sulfasalazine
MeSH Terms: conditions — Alcoholism | interventions — Sulfasalazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sulfasalazine (Experimental): Sulfasalazine 1500 mg
  Interventions: Drug: Sulfasalazine
- Placebo (Placebo Comparator): Placebo capsule x 3 doses 12 hours apart
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sulfasalazine — 500mg capsules of Sulfasalazine x 3 doses 12 hours apart.
  Arms: Sulfasalazine
Drug: Placebo — Placebo capsule x 3 doses 12 hours apart
  Arms: Placebo

SUMMARY:
The overarching objective of this pilot study is to apply both neuroimaging and pharmacogenetic tools to the study of alcohol dependence. This proposed research will provide a mechanistic test of the function of the genetic variation. The specific aims and hypotheses are to test whether Sulfasalazine, as compared to placebo, diminishes blood-oxygen-level dependent (BOLD) response to alcohol cues in the striatum and prefrontal cortex (PFC). To test the hypothesis, we will compare Sulfasalazine treatment with placebo treatment on BOLD difference maps for the contrast alcohol minus control. We will also explore whether specific genetic variations influence this effect. A double-blind, placebo-controlled 2 (Medication: Sulfasalazine 1500 mg vs. placebo control) x 2 (Cue: Alcohol Cue vs. Control cue) within-subjects, crossover design will be used to test the hypothesis that Sulfasalazine reduces the BOLD response in the striatum and prefrontal cortex after exposure to alcohol cues. Twenty alcohol-dependent participants will complete two rounds of the study medication followed by an functional magnetic resonance imaging (fMRI) scan, during which they will complete an alcohol cue-exposure task. The order of the medication condition will be counterbalanced such that subjects will be randomly assigned to receive either Sulfasalazine (1500 mg) in the first session and placebo in the second session one week later (or vice versa). This pilot study will help to determine whether NMDA receptors play a role in cue-elicited activation of key areas of the brain implicated in the development and maintenance of substance use disorders. Furthermore, if Sulfasalazine reduces cue-elicited activation of these brain regions, as hypothesized; this study will lay the groundwork for a larger trial on the efficacy of Sulfasalazine as a treatment for substance use disorders.

DETAILED DESCRIPTION:
The overarching objective of this pilot study is to apply both neuroimaging and pharmacogenetic tools to the study of alcohol dependence. This proposed research will provide a mechanistic test of the function of the genetic variation. The specific aims and hypotheses are to test whether Sulfasalazine, as compared to placebo, diminishes blood-oxygen-level dependent (BOLD) response to alcohol cues in the striatum and prefrontal cortex (PFC). To test the hypothesis, we will compare Sulfasalazine treatment with placebo treatment on BOLD difference maps for the contrast alcohol minus control. We will also explore whether specific genetic variations influence this effect.

Several recent studies support the premise that genetic differences may predict treatment outcomes. In an early study, an A to G single nucleotide polymorphism (SNP; rs1799971) of the mu opiate receptor gene (OPRM1) predicted 12 week abstinence after treatment of alcohol dependence with naltrexone (Oslin et al 2003). The relationship was such that individuals with at least one copy of the G allele demonstrated lower relapse rates and longer time to return to heavy drinking when treated with naltrexone (Oslin et al 2003). These observations were recently replicated and extended in the multisite COMBINE study, such that individuals with the G allele demonstrated superior outcomes after treatment with naltrexone, in combination with medication management (Anton et al 2008). Laboratory studies have suggested that clinical effects may be related to a greater reduction in the acute rewarding effects of alcohol among individuals with the G allele (Ray & Hutchison 2007) and suggest that the mechanism may be related to a blunting of dopamine release in the VTA (Ramchandani et al 2009). In addition, recent studies with other medications (e.g., topiramate, olanzapine) have found that genetic variables predict treatment outcomes (e.g., Hutchison et al 2006; Hutchison 2008; Seneviratne et al 2009). It is important to note that these gene by treatment interactions are not limited to pharmacological treatments, as recent studies have also suggested that genetic variation may predict responses to psychosocial interventions as well (Feldstein Ewing et al 2009; Hutchison et al 2006).

We decided to evaluate the clinical effects of Sulfasalazine because our work to date suggests that genetic variations with downstream function implications for glutamate function, specifically cysteine/glutamate exchange and glutamate transport, are strongly associated with BOLD response in the striatum and prefrontal cortex after exposure to alcohol cues. Sulfasalazine is a medication with a well characterized safety profile that has been used in the treatment of inflammatory bowel disease, including ulcerative colitis and Crohn's disease and several types of arthritis, particularly rheumatoid arthritis for many years. Most recently, it has been suggested that Sulfasalazine may have beneficial effects in the brain, specifically by blocking N-methyl D-aspartate receptor-mediated excitotoxicity resulting in reduced neuronal death (Bo Rum Ryu et al, 2003). This pilot study will help to determine whether NMDA receptors play a role in cue-elicited activation of key areas of the brain implicated in the development and maintenance of substance use disorders. Furthermore, if Sulfasalazine reduces cue-elicited activation of these brain regions, as hypothesized; this study will lay the groundwork for a larger trial on the efficacy of Sulfasalazine as a treatment for substance use disorders.

To that end, a double-blind, placebo-controlled 2 (Medication: Sulfasalazine 1500 mg vs. placebo control) x 2 (Cue: Alcohol Cue vs. Control cue) within-subjects, crossover design will be used to test the hypothesis that Sulfasalazine reduces the BOLD response in the striatum and prefrontal cortex after exposure to alcohol cues. Twenty alcohol-dependent participants will complete two rounds of the study medication followed by an fMRI scan, during which they will complete an alcohol cue-exposure task. The order of the medication condition will be counterbalanced such that subjects will be randomly assigned to receive either Sulfasalazine (1500 mg) in the first session and placebo in the second session one week later (or vice versa).

ELIGIBILITY:
Inclusion Criteria:

* 21-55 years of age with
* Alcohol Dependence

Exclusion Criteria:

* Medical or MRI Contraindications
* Pregnancy
* Allergy to Sulfa medications

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2010-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kent E Hutchison, PhD, Principal Investigator — The Mind Research Network
Locations (1):
- The Mind Research Network, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited in Albuquerque, NM between March 2011 and August 2011.
Pre-assignment Details: 23 participants were recruited; 10 excluded; 13 approved; 1 participant lost to follow-up; 12 participants completed protocol. Of the 12 participants who completed the protocol, each received both interventions: Sulfasalazine first, then placebo, as well as, Placebo first, then Sulfasalazine. Subjects were randomized to intervention order.
Groups:
- Placebo First, Then Sulfasalzine: Placebo x 3 doses 12 hours apart in the first session, followed by a washout period of 7 days, then Sulfasalazine capsule, 500mg, x 3 doses 12 hours apart in the second session (Sulfasalazine 1500mg total)
- Sulfasalazine First, Then Placebo: Sulfasalazine capsule, 500mg, x 3 doses 12 hours apart in the first session (Sulfasalazine 1500mg total) followed by a washout period of 7 days, then Placebo capsule x 3 doses 12 hours apart in the second session.
Period: First Intervention (24 Hours)
Arm/Group | Placebo First, Then Sulfasalzine | Sulfasalazine First, Then Placebo
Started | 6 | 7
Control Cue | 6 | 7
Alcohol Cue | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Placebo First, Then Sulfasalzine | Sulfasalazine First, Then Placebo
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0
Period: Second Intervention (24 Hours)
Arm/Group | Placebo First, Then Sulfasalzine | Sulfasalazine First, Then Placebo
Started | 6 | 7
Control Cue | 6 | 6
Alcohol Cue | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo First, Then Sulfasalazine: Placebo x 3 doses 12 hours apart in the first session, followed by a washout period of 7 days, then Sulfasalazine capsule, 500mg, x 3 doses 12 hours apart in the second session (Sulfasalazine 1500mg total)
- Total: Total of all reporting groups
Arm/Group | Placebo First, Then Sulfasalazine | Sulfasalazine First, Then Placebo | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: % BOLD Response Increase Above Baseline
Description: Test whether Sulfasalazine, as compared to placebo, diminishes blood-oxygen-level dependent (BOLD) response to alcohol cues in the striatum and prefrontal cortex (PFC). BOLD response refers to brain activation in response to the presence of oxygen in a particular part of the brain. To test the hypothesis, we will compare Sulfasalazine treatment with placebo treatment. During the fMRI scan session, participants will be presented with the alcohol cue task. We will compare the difference in BOLD response during the presence of alcohol vs. a novel substance during the alcohol cue task. Outcome data collected during the alcohol cue task will provide us with BOLD response data for each intervention period. We will analyze the outcome data using FSL (Oxford Centre for Functional MRI of the Brain (FMRIB) Software - a collection of functional and structural brain image analysis tools).
Time Frame: Over two weeks
Measure: Mean (Standard Deviation); unit: % BOLD Response increase above baseline
Groups:
- Placebo: Placebo x 3 doses 12 hours apart
- Sulfasalazine: Sulfasalazine capsule, 500mg, x 3 doses 12 hours.
Arm/Group | Placebo | Sulfasalazine
Number analyzed (Participants) | 12 | 12
% BOLD Response increase above baseline
  Control Cue | .106 (.140) | .082 (.156)
  Alcohol Cue | .074 (.167) | .097 (.125)
Statistical Analysis 1: Comparison: Placebo vs Sulfasalazine; Test type: Superiority or Other; p = .05, ANOVA — =0.05 is the actual computed p-value via the ANOVA; The ANOVA is comparing the % increase in BOLD response above baseline during cue presentation (Alcohol vs. Control) b/w placebo & Sulfasalazine

ADVERSE EVENTS:
Arm/Group | Placebo First, Then Sulfasalazine | Sulfasalazine First, Then Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No